CLINICAL TRIAL: NCT05281536
Title: Effects of Trunk Postural Change on CO2 Removal Efficiency in ARDS Patients: Quasi-experimental Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica las Condes, Chile (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: E012021
Record Dates: First submitted 2022-03-07; First posted 2022-03-16 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: ARDS
Keywords: Trunk Inclination; Postural change; Dead space; ARDS
MeSH Terms: interventions — Supine Position

STUDY DESIGN:
Intervention Model Description: The intervention will be a postural change from 45° to 10° in a semi-recumbent position of ARDS patients connected to mechanical ventilation.
Masking Description: Data obtained for mechanical ventilation, volumetric capnography, and electric impedance tomography will be download by different investigators when all patients have been recruited.
  The results will be analyzed by statisticians, who will not know the participant's identification
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Postural Changes from 45° to 10° in supine decubitus (Experimental): Postural changes from 45° to 10° in supine decubitus Three times of 60 minutes each step before (45°, baseline) - during (10°, intervention) - after (45°, control)
  Interventions: Other: Ppostural change from 45° to 10° in supine position

INTERVENTIONS:
Other: Ppostural change from 45° to 10° in supine position — The intervention will be a postural change from 45° to 10° in a semi-recumbent position of ARDS patients connected to mechanical ventilation.

SUMMARY:
OBJECTIVES: The trunk inclination from semirecumbent to lying supine improves lung mechanics and reduces end-expiratory lung volume in Acute Respiratory Distress Syndrome (ARDS) patients. Besides, it can improve the ventilatory ratio and PaCO2, although the effects and mechanisms are not entirely elucidated. Therefore, this study aimed to evaluate the effects of trunk tilt from 45° to 10° on CO2 removal efficiency.

DESIGN: Quasi-experimental study. SETTING: A medical ICU in Chile. PATIENTS: Twenty-two patients with ARDS. INTERVENTION: Patients in pressure-controlled ventilation underwent three 60-minute steps in which trunk inclination was changed from 45° (baseline) to 10° (intervention) and back to 45° (control) in the last step. Respiratory mechanics, arterial blood gas analysis, dead space by volumetric capnography, and electrical impedance tomography were recorded.

DETAILED DESCRIPTION:
The role of trunk inclination in the lying position and its physiological effects have been extensively studied in patients with acute respiratory distress syndrome (ARDS).

Consistently, driving pressure and respiratory system compliance (CRS) increase has been found when bed angulation is increased at 40 - 45 degrees. Besides, most patients in the semi-recumbent position rising end-expiratory lung volume (EELV) and oxygenation. These findings continue to raise questions regarding the physiological mechanisms underlying these effects.

On the other side, changing trunk tilt to zero degrees in patients with COVID-19 related ARDS reduced the ventilatory ratio and partial pressure of carbon dioxide (PaCO2). In addition, when patients were placed in a lying-flat position at 0°, the driving pressure and lung compliance declined, generating lower energy applied to the lung. This way, an alveolar overdistention reduction could explain the improvement in the kinetics of CO2 but is not fully elucidated, mainly due to the short evaluation period and the low accuracy of the ventilatory ratio to measure the lung efficiency to exhale CO2. It should be noted that one of the best ways to assess ventilatory efficiency physiologically is with volumetric capnography (8), but this technology has never been used when chest inclination changes in ARDS patients.

Thus, we hypothesized that changes in trunk inclination to a lying-flat position in ARDS patients connected to mechanical ventilation would improve CO2 removal efficiency. Therefore, the primary objective of this study was to assess the effects of postural change from 45° to 10° bed tilt on CO2 exhaled per minute (VCO2), Bohr's dead space (VDBohr/VT) and PaCO2. The secondary objective was to evaluate the lung volume effects and the ventilation distribution in the different lung regions.

Study steps:

step I: Baseline conditions. Patient in the semi-recumbent position at 45° head-up, and lower extremities parallel to the floor.

step II: Intervention phase with a trunk postural change at 10° in lying supine position.

step III: Control phase with a return to the semi-recumbent position at 45° head-up.

Five minutes before each step, PaCO2, and partial pressure of arterial oxygen over the fraction of inspired oxygen (PaO2/FIO2) were recorded. Both tidal volume (VT), volumetric capnography and Electrical impedance tomography (EIT) variables were analyzed offline using the mean value of the last 20 breaths of the last three minutes of each step. Haemodynamic variables and pulse oximetry were continuously monitored (Multiparameter Spacelabs 91393 Xprezzon®).

Security procedure:

Therapeutic interventions were kept strictly unchanged during all evaluation periods. The following criteria were predefined to interrupt the study protocol if required: desaturation corresponding to a drop of more than 10% of baseline oxygen saturation value; drop in mean arterial pressure of more than 20% of baseline value or heart rate increase of more than 20 % of baseline values.

Primary outcomes:

VDBohr/VT and PaCO2 reduction at 60 minutes of trunk change to 10° concerning the body position in basal conditions of 45°.

Statistical analysis:

Different assumptions were made for a repeated sample study. We considered as clinically significant effect, a mean reduction of 5 mmHg with a standard deviation of ± 3 mmHg of PaCO2 with a power of 90% and a probability of type I error of 0.01. Based on these assumptions, the sample size was 22 participants.

The Shapiro-Wilk test was performed to determine the distribution of continuous variables while homoscedasticity was tested using the Levene test. According to their distribution, continuous variables were expressed as mean and standard deviation or median and interquartile range. Parametric versus non-parametric tests were decided according to the data distribution and whether the assumption of normality was met. Continuous variables were analyzed by ANOVA for repeat measure, or the Friedman test was applied, as appropriate. Bonferroni and Dunn's post hoc were used for the comparison between step II-step I, step III-step I and step III-step II, respectively.

T-test was used to measure the median difference and 95% confidence interval (95% CI) between step I and step II. Wilcoxon rank test was performed to evaluate changes in ventral or dorsal end-expiratory lung impedance (EELI) and tidal variation of impedance (VTI) from 45 to 10 degrees.

A two-tailed p-value less than 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18 years old
2. Admitted to Intensive Care with mild, moderate, or severe ARDS according to the Berlin classification
3. Less than 72 hours of connection to mechanical ventilation.
4. Depth Sedation-analgesia.
5. Acceptance by the legal representative to participate in the study.

Exclusion Criteria:

1. Pleural tube - bronchopulmonary fistula.
2. Prone position
3. Hypovolemic shock with active bleeding.
4. Intracranial hypertension.
5. Gastric residue greater than 300 ml in the last 6 hours
6. Hemodynamic instability that requires a progressive increase in the dose of vasopressors
7. Temperature variations greater than 0.5 ° C in the last 2 hours
8. Acute heart failure
9. Chronic respiratory disease (FEV1 <50% predicted).
10. Patients who do not have an arterial line.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Changes in PaCO2 | 60 minutes each phase
  Determine the effects of postural changes from 45° to 10° on PaCO2
Changes in Bohr's dead-space | 60 minutes each phase
  Determine the effects of postural changes from 45° to 10° on Bohr's dead-space

CONTACTS AND LOCATIONS:
Overall Officials: Martín Benites, MD, Principal Investigator — Clínica Las Condes
Locations (2):
- Chile (2):
  - Clínica Las Condes, Santiago, Santiago Metropolitan
  - Martín Hernán Benites, Santiago, Santiago Metropolitan

IPD SHARING:
Plan to Share IPD: No
I would have to request authorization from the institutional ethics committee to provide the information.
  Should you need any further information, please do not hesitate to contact me. benitesmartinh@gmail.com

REFERENCES:
- [Background] Marrazzo F, Spina S, Forlini C, Guarnieri M, Giudici R, Bassi G, Bastia L, Bottiroli M, Fumagalli R, Langer T. Effects of Trunk Inclination on Respiratory Mechanics in Patients with COVID-19-associated Acute Respiratory Distress Syndrome: Let's Always Report the Angle! Am J Respir Crit Care Med. 2022 Mar 1;205(5):582-584. doi: 10.1164/rccm.202110-2360LE. No abstract available. PMID 34982652
- [Result] Tusman G, Gogniat E, Bohm SH, Scandurra A, Suarez-Sipmann F, Torroba A, Casella F, Giannasi S, Roman ES. Reference values for volumetric capnography-derived non-invasive parameters in healthy individuals. J Clin Monit Comput. 2013 Jun;27(3):281-8. doi: 10.1007/s10877-013-9433-x. Epub 2013 Feb 7. PMID 23389294
- [Result] Mentzelopoulos SD, Roussos C, Zakynthinos SG. Static pressure volume curves and body posture in acute respiratory failure. Intensive Care Med. 2005 Dec;31(12):1683-92. doi: 10.1007/s00134-005-2838-3. Epub 2005 Oct 26. PMID 16249926
- [Result] Rehder K. Postural changes in respiratory function. Acta Anaesthesiol Scand Suppl. 1998;113:13-6. doi: 10.1111/j.1399-6576.1998.tb04980.x. PMID 9932113